CLINICAL TRIAL: NCT04071704
Title: Incorporating the Patient Voice in Sarcoma Research: How Can we Assess Health-related Quality of Life in This Heterogeneous Group of Patients?
Brief Title: Assessing Health-related Quality of Life in Sarcoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Radboud University Medical Center (Other); Leiden University Medical Center (Other); Centre Leon Berard (Other); University Hospital Carl Gustav Carus (Other); Heidelberg University (Other); Johannes Gutenberg University Mainz (Other); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); National Cancer Institute, Naples (Other); Maria Sklodowska-Curie National Research Institute of Oncology (Other); Hospital San Carlos, Madrid (Other); Royal Marsden NHS Foundation Trust (Other); Beatson West of Scotland Cancer Centre (Unknown); University Hospital Southampton NHS Foundation Trust (Other); Royal National Orthopaedic Hospital NHS Trust (Other); Bank of Cyprus Oncology Centre (Other); Institut Català d'Oncologia (Other); University of Adelaide (Other); King Hussein Cancer Center (Other); Oslo University Hospital (Other); Erasmus Medical Center (Other); University Medical Center Groningen (Other); Centre Oscar Lambret (Other); Aretaieio Hospital (Other); Hospital Universitario Fundación Jiménez Díaz (Other); The Christie NHS Foundation Trust (Other); Ain Shams University (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other); Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: EORTC-1749
Record Dates: First submitted 2019-08-08; First posted 2019-08-28 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Sarcoma
Keywords: health-related quality of life; life satisfaction; treatment-related effects; quality of life measure
MeSH Terms: conditions — Sarcoma; Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients who have been or are being treated for sarcoma.
- Health care professionals: Health care professionals with extensive experience in sarcoma care (medical oncologists, radiation oncologists, surgical oncologists, orthopaedic surgeons, nurse specialists, psychologists, physiotherapists)

SUMMARY:
Although the clinical effectiveness of sarcoma treatment has improved, long-lasting and cumulative treatment side-effects may often detract from the overall marginal advantage. Information only on survival is insufficient to determine the net clinical benefit of a treatment. It is important to assess treatment effectiveness both in terms of objective outcomes (e.g., response, recurrence and survival) and in terms of subjective patient reported outcomes (PROs), objective functional outcomes including health-related quality of life (HRQoL).

Previous studies have predominantly used generic HRQoL instruments, which cover some relevant issues but do not capture all the unique experiences of patients with sarcoma, and thus lack content validity. A sarcoma-specific questionnaire should be able to detect, with more sensitivity, side-effects, symptoms and problems with function that are particularly relevant to patients with sarcoma. To date , there is no specific sarcoma HRQoL instrument available; and, given the heterogeneity of the disease in terms of subtype, location, age and treatment, the development of such an instrument may be challenging.

The aim of this collaborative project between the EORTC Quality of Life Group (QLG) and the EORTC Soft Tissue and Bone Sarcoma Group (STBSG) is to raise the standard of HRQoL measurement in patients with sarcoma. An important question remains to be answered: Is it possible to develop one PROs questionnaire covering HRQoL issues that are relevant to all adult patients with sarcoma, or are the HRQoL issues related to the different localization / treatment sufficiently different to warrant the creation of separate item lists selected from the EORTC QLG Item Library?

DETAILED DESCRIPTION:
The investigators will follow the EORTC QLG questionnaire development guidelines. First, a computerized search of the academic literature will be performed to identify all relevant HRQoL issues for and existing HRQoL questionnaires currently used among patients with sarcoma. In parallel, semi-structured interviews will be conducted worldwide with patients with sarcoma(N=179) and health care professionals (HCPs; N=35; phase 1a). The patient sample will be stratified to capture diversity across the sarcoma population tumour location (extremities, axial, head and neck, thorax, retroperitoneal/intra-abdominal and gynecological), stage (localized vs. metastatic disease ) and type or lines of treatment .

This list of HRQoL issues generated by the a) literature search, b) relevant items from the Item Library, and c) semi-structured patient and HCP interviews, and will be consolidated into a comprehensive list of issues for all languages of collaborating countries.

In phase 1b, the new list of HRQoL issues will be presented to another group of patients with sarcoma(N=475) and HCPs (N=72). Patients and HCPs will be asked to rate the HRQoL issues on relevance (4point Likert scale) and to prioritize the 10 most important issues.

ELIGIBILITY:
Inclusion Criteria:

* Age at diagnosis 18 years or older
* Having a confirmed diagnosis of sarcoma

Exclusion Criteria:

* Having any psychiatric condition or cognitive impairment that would hamper participation in interview/completion of self-reported questionnaires.
* Patients with a Gastrointestinal Stroma Tumour (GIST) diagnosis, as they are quite unique in terms of type of disease and treatment.
* Patients with Kaposi sarcoma, as this disease occurs quite often in people with AIDS
* Patients with Carcinosarcoma as this disease is generally seen as a carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with sarcoma, with all stages of disease. The primary types of treatments to be included, depending on sarcoma subtype, are chemotherapy/targeted therapy, radiotherapy, surgery, or a combination of these.
Sampling Method: Non-Probability Sample
Enrollment: 689 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
a framework for a HRQoL measure for patients with sarcoma | 1 week (and for several issues 4 weeks according to EORTC questionnaire guidelines)
  the framework will outline which strategy to adopt for HRQoL in patients with sarcoma: the EORTC Quality of Life Questionnaire (QLQ)-C30 + one sarcoma module; EORTC QLQ-C30 + one sarcoma module + an item list; EORTC QLQ-C30 + item list.
  This will be based on analysis of the interview data (patients and HCPs) and the relevance of certain HRQoL rated by patients and health care professionals and possible identification of certain subgroups (according to tumour localization, type of sarcoma, disease stage and treatment).

SECONDARY OUTCOMES:
an exhaustive list of all HRQoL issues relevant to sarcoma patients | 1 week (and for several issues 4 weeks according to EORTC questionnaire guidelines)
  based on a literature review, analysis of interviews with patients and health care professionals we will create an exhaustive list of all HRQoL issues relevant to sarcoma patients.
the coverage of issues/items already available in the EORTC Item Library | 1 week (and for several issues 4 weeks according to EORTC questionnaire guidelines)
  the interview data and rating of HRQoL issues will be used to determine the overage of issues/ items in the EORTC Item Library and how the Item Library can be optimally used for the HRQoL measure for patients with sarcoma.
the proportion of patients in subgroups rating issues/items as relevant | 1 week (and for several issues 4 weeks according to EORTC questionnaire guidelines)
  In order to determine if issues are sarcoma-generic or dependent of sarcoma localization, sarcoma subtype, disease stage or treatment we will analyze the proportion of patients in each subgroup rating HRQoL issues or items as relevant

CONTACTS AND LOCATIONS:
Overall Officials: Olga Husson, PhD, Principal Investigator — The Netherlands Cancer Institute; Winette van der Graaf, PhD, MD, Principal Investigator — The Netherlands Cancer Institute
Locations (3):
- Germany (2):
  - University Hospital Carl Gustav Carus, Dresden
  - Johannes Gutenberg University Mainz, Mainz
- Kiing Hussein Cancer Centre, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] den Hollander D, Lidington E, Singer S, Sodergren SC, Salah S, Fiore M, Benson C, Desar IME, Burgers VWG, Husson O, van der Graaf WTA. 'I thought I had fibroids, and now I don't': a mixed method study on health-related quality of life in uterine sarcoma patients. Health Qual Life Outcomes. 2022 Apr 20;20(1):65. doi: 10.1186/s12955-022-01971-5. PMID 35443673
- [Derived] den Hollander D, Fiore M, Martin-Broto J, Kasper B, Casado Herraez A, Kulis D, Nixon I, Sodergren SC, Eichler M, van Houdt WJ, Desar IME, Ray-Coquard I, Piccinin C, Kosela-Paterczyk H, Miah A, Hentschel L, Singer S, Wilson R, van der Graaf WTA, Husson O. Incorporating the Patient Voice in Sarcoma Research: How Can We Assess Health-Related Quality of Life in This Heterogeneous Group of Patients? A Study Protocol. Cancers (Basel). 2020 Dec 22;13(1):1. doi: 10.3390/cancers13010001. PMID 33561018